CLINICAL TRIAL: NCT06120907
Title: Swiss Itch Registry (SWITCHR) - A Prospective Registry to Collect Data of Patients With Chronic Pruritus
Brief Title: Swiss Itch Registry
Acronym: SWITCHR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00310; th21Mueller
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Pruritus
Keywords: Itch; Chronic pruritus (CP)
MeSH Terms: conditions — Pruritus | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Biospecimen Retention: Samples With DNA — Blood plasma; Skin punch biopsies. All biological material will be integrated and stored in -80̊ C freezer in a restricted area of the biobank of the Department of Dermatology of the University of Basel according to the current version of the biobank regulation for an indefinite duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — The data include phenotypic data, treatments administered, response to treatment, Three-dimensional total body images, biopsies and blood plasma.

SUMMARY:
This project is to develop a national registry for CP patients. Patients admitted to this registry will be examined and documented with PROs, physician-based assessments, blood tests, 3D photodocumentation and, if indicated, by skin biopsies, neurophysiological testing and radiological imaging at defined timepoints. The data collection will allow deepened insights into patient needs, different mechanisms and courses of pruritic conditions, treatment outcomes and treatment-related safety issues. In addition, the collection of clinical, biological and image-based data may be used for retrospective analyses.

DETAILED DESCRIPTION:
Pruritus (synonymous "itch") is the commonest skin-related symptom caused by numerous dermatological and non-dermatological conditions. Chronic pruritus (CP) defined by a duration of > 6 weeks is associated with significantly impaired quality of life and high socio-economic burden. At present, a data registry to monitor and compare clinical presentation, treatment outcomes and safety issues of these patients is lacking in Switzerland. The implementation of the SWITCHR could help to i.) improve medical care of CP patients, ii.) allow standardised comparison of different pruritic conditions as well as national data with international CP populations and iii.) raise the awareness for CP in general practitioners, health care institutions, national public health authorities and pharmaceutical companies within Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years.
* Written informed consent of the patient.
* Diagnosis of CP irrespective of the International Forum for the Study of Itch (IFSI) group (I-III) and/or underlying cause (according to the judgment of the investigator).
* A Numerical Rating Scale (NRS) score of min. ≥ 4 within the last 7 days.
* Sufficient language skills (in the languages which the patient information and the consent form is available) to provide informed consent.

Exclusion Criteria:

* Any medical or psychological condition in the treating physician's opinion, which may prevent the patient in registry participation
* Lack of informed consent for registry participation.
* Refusal to complete Patient Reported Outcomes (PROs)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited by consecutive ongoing recruitment in the investigators' clinical practice during 10 years.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2033-10 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Change in Dermatology Life Quality Index (DLQI) | up to 60 months
  The Dermatology Life Quality Index (DLQI) consists of 10 questions concerning patient's perception of the impact of skin diseases on different aspects of their health-related QoL over the last week. The DLQI evaluates the impact of the patient's skin disease on daily activities, leisure, work and personal relationships. DLQI score 0-1 = no effect at all on patient's life DLQI score of 2-5 = small effect on patient's life, DLQI score of 6-10 = moderate effect on patient's life, DLQI score of 11-20 = very large effect on patient's life, DLQI score of 21-30 = extremely large effect on patient's life.
Change in ItchyQoL questionnaire | up to 60 months
  The ItchyQoL is a questionnaire to measure the quality of life in CP patients. It is composed of 22 items regarding symptoms, functions, emotions and self-perception. Each of the questions is scored 1-5 (1:never; 2: rarely; 3: sometimes; 4: often; 5: all of the time) withthe sum forming the raw ItchyQol score with a range of 22-110.
Change in NeuroDerm questionnaire | up to 60 months
  This questionnaire comprises questions and descriptions deemed to be clinically relevant for chronic pruritus: It consists of a general part and special modules such as beginning and course, topographical distribution, influencing factors, intensity, quality of CP.
Change in Itch Controlled Days (ICD) Questionnaire | up to 60 months
  This questionnaire consists of eight items addressing itch intensity, scratching behaviour, itch-related sleep disturbance and temporal aspects of feeling itchy.
Change in Dynamic Pruritus Score (DPS) | up to 60 months
  This score compares the reduction in the current level of pruritus with a defined point earlier in time. It is comprised of a horizontal line measuring itch improvement via 11 marks on a scale, each labelled with both a numerical and verbal description.
Change in Regensburg Insomnia Scale (RIS) | up to 60 months
  This 10-item rating scale is designed for the assessment of psychophysiological insomnia and is composed of 10 different sections addressing latency, duration, continuity, depth of sleep, experience of sleepless nights, sleep-related thoughts or fear, and use of sleep medication. Total scores range from 0 to 40 points with higher scores indicative of more cognitive, behavioural, and emotional difficulties consistent with psychophysiological insomnia. Scores from 0-12 are considered normal and scores above the cutoff (13+) are indicative of symptoms consistant with psychophysiological insomnia that warrant further investigation.
Change in Itch-related patient's drawing | up to 60 months
  Patients (on a voluntary basis) draw their itch-related perception, emotions, concerns, wishes and desires in a 10- minutes sketch. Drawings of CP patients usually contain additional diagnostic information not captured in usual history taking and might also be helpful to discuss treatment strategies in an "imaged-based" manner.
Change in the Eight-item Patient Health Questionnaire (PHQ-8) | up to 60 months
  The Eight-item Patient Health Questionnaire (PHQ-8) is a tool for the screening of depression (presence and severity). PHQ-8 questions refer to the last two weeks, addressing the level of interest in doing things, feeling down or depressed, difficulty with sleeping, energy levels, eating habits, self-perception, ability to concentrate, speed of functioning and thoughts of suicide. The score range is 0 to 27 (0-4 = none- minimal, 5-9 = mild, 10-14 = moderate, 15-19 = moderate severe, 20-27 = severe)
Change in the Somatic Symptom Scale-8 (SSS-8) | up to 60 months
  The Somatic Symptom Scale-8 (SSS-8) is a brief version of the Patient Health Questionnaire-15 (PHQ-15) used to assess somatic symptom burden during the last two weeks. It measures the perceived burden of common somatic symptoms. (Score 0-3 = Severity: No to minimal. Score: 16 - 32 = Severity: Very high)
Change in the Somatic Symptom Disorder - B Criteria Scale (SSD-12) | up to 60 months
  The Somatic Symptom Disorder - B Criteria Scale (SSD-12) is a brief self-report questionnaire used to assess the patient's perception of symptom-related thoughts, feelings, and behaviors during the last 30 days. The SSD-12 consists of 12 questions and measures three psychological sub-criteria (cognitive, affective, and behavioral) with scores between 0 and 4 (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = very often)
Change in the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | up to 60 months
  The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) consists of 12 questions, covers 6 domains of functioning (cognition, mobility, self-care, getting along, life activities, participation) and asks about difficulties during the last 30 days due to diseases or other health problems. The scores assigned to each of the items-"none" (1), "mild" (2), "moderate" (3), "severe" (4), and "extreme" (5)-are summed.
Change in the Generalized Anxiety Disorder 7 (GAD-7) | up to 60 months
  The Generalized Anxiety Disorder 7 (GAD-7) is a self- reported questionnaire for screening and assessment of the severity of generalized anxiety disorder (GAD). It consists of 7 questions including nervousness, inability to stop worrying, excessive worry, restlessness, difficulty in relaxing, easy irritation and fear of something awful happening. Each item is rated from 0-15+ ((0-4 = No to Low risk, 5-9 = mild, 10-14 = moderate, 15+ = severe)
Change in the SCORing Atopic Dermatitis (SCORAD) | up to 60 months
  SCORing Atopic Dermatitis (SCORAD) is a clinical tool for assessing the extent (A: according to the rule of nines; 20% of the score), the intensity composed of six items (B: erythema, oedema/papules, effect of scratching, oozing/crust formation, lichenification and dryness; 60% of the score; each item has four grades: 0, 1, 2, 3) and subjective symptoms (C: itch, sleeplessness; 20% of the score) which are rated on a 0-10 VAS.
Change in the Eczema Area and Severity Index (EASI) | up to 60 months
  The Eczema Area and Severity Index (EASI) is a tool used to measure the extent (area) and severity of atopic eczema. Inflamed areas of four body regions (head and neck, trunk, upper limbs and lower limbs) are assessed. The area score ranging from 0-6 is the percentage of skin affected by eczema for each body region (0 = no active eczema in this region, 1= 1-9%, 2 = 10-29%, 3 = 30-49%, 4 = 50-69%, 5 = 70-89%, 6 = 90-100%: the entire region is affected by eczema).
Change in the Psoriasis Area and Severity Index (PASI) | up to 60 months
  The Psoriasis Area and Severity Index (PASI) is a composite variable used to assess the severity of Psoriasis. The PASI evaluates the area of psoriatic involvement in 4 main areas (head, trunk, upper and lower extremities) and the severity of the psoriatic lesions with respect to three target symptoms: erythema, infiltration and desquamation, each to be rated on a scale from 0-4.
Change in the Physician Global Assessment (PGA) | up to 60 months
  The Physician Global Assessment (PGA) relies on clinical assessment of the patient's skin presentation. The investigator (or qualified site personnel) scores the erythema, pustules, and scaling of all lesions on a scale from 0 to 4. Each component is graded separately, the average is calculated, and the final PGA is determined based on this composite score. A lower score indicates a lower severity, with 0 being clear and 1 being almost clear.
Change in the Investigator's Global Assessment of Chronic Prurigo (IGA-CPG) | up to 60 months
  The Investigator's Global Assessment of Chronic Prurigo is designed to categorize the stage and activity of chronic prurigo and prurigo nodularis on scores from 0-4 each.
Change in Quantitative Sensory Testing (QST) | up to 60 months
  QST measures the detection threshold of accurately calibrated sensory stimuli (i.e. touch, vibration, thermosensation, pain). It quantifies individual sensory perceptions using direct patient feedback. Subject values are compared to normal data to determine whether the subject has a deficit in any modality.
Change in skin surface by 3DSkin imaging (Vectra®) | up to 60 months
  The Vectra whole-body scanner is a high-definition 3D-visual documentation creating a 3D avatar, capturing nearly the entire skin surface. It monitors itch-related primary and secondary skin lesions, scratching patterns and treatment responses.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mueller, PD Dr. med., Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland